CLINICAL TRIAL: NCT04932031
Title: Systemic Assessment of CIPN Risk Using Molecular Aging Trajectories
Brief Title: Risk Prediction of Taxane Chemotherapy-Induced Peripheral Neuropathy
Acronym: SENSE
Status: Terminated | Type: Observational
Why Stopped: under enrollment for primary endpoint analysis
Sponsor: Sapere Bio (Industry)
Collaborators: National Institute on Aging (NIA) (NIH); University of North Carolina (Other); University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Other Study IDs: SB-2101
Record Dates: First submitted 2021-06-12; First posted 2021-06-18 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Breast Cancer; Chemotherapy-induced Peripheral Neuropathy; Aging
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood an plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Adult females with newly diagnosed early-stage (stages I III) non-metastatic breast cancer receiving neoadjuvant or adjuvant chemotherapy that includes paclitaxel or docetaxel

SUMMARY:
This is an observational study to discover risk factors of chemotherapy-induced peripheral neuropathy (CIPN) in 350 patients with early stage breast cancer undergoing taxane-based chemotherapy at two main sites (University of North Carolina at Chapel Hill (UNC) Hospital, including Rex Hospital, and the University of Alabama at Birmingham (UAB) Hospital). The primary purpose of this study to explore patient- and procedure-based variables that identify patients at risk for developing CIPN during chemotherapy.

DETAILED DESCRIPTION:
Chemotherapy-induced peripheral neuropathy is common and provokes pain, poor QoL, and loss of independence, as well as increases the risk of falls and opioid addiction. Beyond the inciting agents, risk factors for CIPN are not understood or systematically evaluated in clinical practice, precluding prevention. Therefore, a clinical decision tool to predict an individual patient's risk of neuropathy remains a critical unmet need. A diagnostic test that predicts CIPN risk in this clinical context would provide an essential clinical-decision tool to guide treatment and post-treatment care in breast cancer, prevent CIPN occurrence, and improve patient outcomes.

Investigators' pilot data uncovered a strong association between cellular senescence and CIPN. In this prospective, observational study of participants with early-stage breast cancer, the investigators will assess the contribution of senescence and clinical variables. The investigators will determine the ability of these factors to identify patients at risk for CIPN during chemotherapy and up to one year after the last dose of taxane-based chemotherapy. This study will employ both patient- and clinician reported CIPN scoring systems.

ELIGIBILITY:
Inclusion Criteria:

Study participants must meet all of the following inclusion criteria to participate in the study:

* Adult female study participants (≥18 years) with newly diagnosed early-stage (stages I III) non-metastatic breast cancer receiving neoadjuvant or adjuvant chemotherapy that includes paclitaxel or docetaxel
* Study participants must be capable and willing to provide informed consent, and be willing and able to complete the study questionnaires during the study

Exclusion Criteria:

Study participants who fulfill any of the following criteria will be excluded:

* Patients with metastatic breast cancer
* History of other cancers (except squamous and basal cell carcinoma)
* Autoimmune disorders
* Presence of major active infection for which antibiotics and/or antivirals are prescribed within the last 14 days (chronic or acute, eg, sepsis, HIV, pneumonia, active COVID infection)
* Pregnant women
* Participation in an additional study at the time of enrollment where the intervention could potentially alter CIPN risk (unless in the control arm)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — enrollment is based on the biological sex due to the nature of the disease
Study Population: Adult female study participants (≥18 years) with newly diagnosed early-stage (stages I III) non-metastatic breast cancer receiving neoadjuvant or adjuvant chemotherapy that includes paclitaxel or docetaxel
Sampling Method: Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2022-05-25 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Change between baseline and the peak EORTC QLQ CIPN20 score during chemotherapy (continuous) | 12 weeks
  EORTC QLQ CIPN20

SECONDARY OUTCOMES:
Incidence of grade 2 or higher CTCAE-CIPN during chemotherapy (binary) | 12 weeks
  CTCAE-CIPN
Dose reduction or discontinuation of chemotherapy (<85% of planned total dose delivered) (binary) | 12 weeks
  dose reduction or discontinuation
Dose reduction or discontinuation of the taxane portion of the chemotherapy, if administered separately from the rest of the chemotherapy agents (<85% of planned total dose delivered) (binary) | 12 weeks
  dose reduction or discontinuation
Change between baseline and the EORTC QLQ-CIPN20 score at one year after the last taxane-based chemotherapy dose (continuous) | 1 year
  EORTC QLQ-CIPN20
Presence of CIPN at one year after the last taxane based chemotherapy dose that is an EORTC QLQ-CIPN20 score of 3 points or higher than baseline (binary) | 1 year
  EORTC QLQ-CIPN20
Presence of grade 2 or higher CTCAE-CIPN at one year after the last taxane-based chemotherapy dose (binary) | 1 year
  CTCAE-CIPN

OTHER OUTCOMES:
Calculation of total chemotherapy dose delivered using a longitudinal cumulative dose of chemotherapy formula | 12 weeks
  Longitudinal cumulative dose of chemotherapy formula

CONTACTS AND LOCATIONS:
Overall Officials: Natalia Mitin, PhD, Principal Investigator — Sapere Bio
Locations (2):
- United States (2):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - UNC Hospitals Adult Oncology Clinics, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: No